CLINICAL TRIAL: NCT00697086
Title: Efficacy and Safety of Dronedarone for the Control of Ventricular Rate During Atrial Fibrillation (ERATO)
Brief Title: European Study of Dronedarone in Atrial Fibrillation
Acronym: ERATO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4508; SR33589
Record Dates: First submitted 2008-06-12; First posted 2008-06-13 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Atrial Fibrillation
Keywords: Heart disease
MeSH Terms: conditions — Atrial Fibrillation; Heart Diseases | interventions — Dronedarone

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Dronedarone (SR33589)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronedarone (SR33589)
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy of dronedarone for the control of ventricular rate at rest and during exercise in patients with atrial fibrillation (AF) and to assess the tolerability of dronedarone in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic permanent AF (>6 months) for which cardioversion is not considered and resting ventricular rate > or equal 80 bpm at screening measured on a 6-seconds rhythm strip,

Exclusion Criteria:

* Unstable angina pectoris, recent myocardial infarction or history of torsades de pointes
* Third degree atrioventricular block at the screening ECG or significant sinus node disease without a permanent pacemaker implanted
* Clinically overt congestive heart failure at randomization
* Patients treated with amiodarone, other antiarrhythmic drugs or previous participation in this trial or in other dronedarone trials or taking an investigational drug
* Clinically relevant haematologic, hepatic, gastro-intestinal, renal, pulmonary, endocrinologic or psychiatric disease
* Pregnant and/or breastfeeding women or women of child-bearing potential with no adequate birth control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2002-08; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean ventricular rate at rest and during exercise | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (9):
- Sanofi-aventis Administrative Office, Diegem, Belgium
- Sanofi-aventis Administrative Office, Prague, Czechia
- Sanofi-aventis Administrative Office, Paris, France
- Sanofi-aventis Administrative Office, Milan, Italy
- Sanofi-aventis Administrative Office, Gouda, Netherlands
- Sanofi-aventis Administrative Office, Warsaw, Poland
- Sanofi-aventis Administrative Office, Barcelona, Spain
- Sanofi-aventis Administrative Office, Bromma, Sweden
- Sanofi-aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Result] Davy JM, Herold M, Hoglund C, Timmermans A, Alings A, Radzik D, Van Kempen L; ERATO Study Investigators. Dronedarone for the control of ventricular rate in permanent atrial fibrillation: the Efficacy and safety of dRonedArone for the cOntrol of ventricular rate during atrial fibrillation (ERATO) study. Am Heart J. 2008 Sep;156(3):527.e1-9. doi: 10.1016/j.ahj.2008.06.010. PMID 18760136
- See also: Related Info — http://www.sanofi-aventis.com